CLINICAL TRIAL: NCT03558386
Title: A Multi-Center, Phase II Cross-sectional Study Investigating Quality of Life in Older vs. Younger Adult Patients Undergoing Allogeneic Hematopoietic Cell Transplantation for Myelodysplastic Syndromes: a Companion Study to the CIBMTR 10-CMSMDS-1-Approved Expanded Access Study
Brief Title: Study of Quality of Life in Older vs. Younger Adult Patients Undergoing Allogeneic Hematopoietic Cell Transplantation for Myelodysplastic Syndromes
Status: Completed | Type: Observational
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Other Study IDs: 17-ePRO
Record Dates: First submitted 2018-04-10; First posted 2018-06-15 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Myelodysplastic Syndromes; Hematopoietic Cell Transplant
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients between 55-64 years of age: Patients between 55-64 years who have had a transplant at the following time points:
  * 6 months to 1 year ago
  * 1 year to 3 years ago
  * 3 years ago or more
  Interventions: Behavioral: ePRO survey
- Patients 65+ years of age: Patients 65+ years of age who have had a transplant at the following time points:
  * 6 months to 1 year ago
  * 1 year to 3 years ago
  * 3 years ago or more
  Interventions: Behavioral: ePRO survey

INTERVENTIONS:
Behavioral: ePRO survey — An electronic patient reported outcomes survey will be completed by the patient.

SUMMARY:
This is a multi-center, Phase II, cross-sectional study comparing quality of life (QOL) as assessed by patient-reported outcomes (PROs) in older (≥65 years) adults vs younger (55-64 years) undergoing allogeneic hematopoietic cell transplantation (HCT) for myelodysplastic syndromes (MDS).

DETAILED DESCRIPTION:
Transplant recipients who have met the inclusion and exclusion criteria and from participating study sites will be asked to complete an online consent and survey for the study. This survey is the patient-reported outcomes survey and will be used to assess quality of life. The survey results will then be compared by age group and by time post transplant, between 6 months and a year post transplant, 1 year to 3 years post transplant, and 3 years or more post transplant.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate on this study, an individual must meet all of the following criteria:

1. Underwent an allogeneic HCT for MDS on the 10-CMSMDS-1 protocol
2. Prior consent to research and future contact by the CIBMTR
3. Ability to provide RCI BMT protocol 17-ePRO signed and dated informed consent form (ICF)
4. Age ≥55 years at time of transplant
5. Fluent in English or Spanish
6. Greater than 6 months post-HCT

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation on this study.

1. No access to an internet browser or email account
2. Within 6 months of first HCT for MDS on the 10-CMSMDS-1 protocol

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects previously enrolled on the 10-CMSMDS-1 protocol at participating centers will be assessed for eligibility into this protocol. Those meeting inclusion and exclusion criteria and consenting to participate will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Long-term post-HCT QOL (in particular physical function and fatigue) for transplant recipients ≥65 years old to those 55-64 years old. | Those completing the assessment at one timepoint 6 months-1 year post-HCT, Those completing the assessment at one timepoint 1 year - 3 years post-HCT, Those completing the assessment at one timepoint Greater than 3 years post-HCT
  The primary objective is to compare the change in long-term post-HCT QOL (in particular physical function and fatigue) for transplant recipients ≥65 years old to those 55-64 years old as measured by the assessment and when the assessment occurred at a post-HCT timepoint.

SECONDARY OUTCOMES:
Domain-specific QOL scores by age group as assessed by PROMIS measures. | 6 months-1 year post-HCT, 1 year - 3 years post-HCT, 3 years+ post-HCT
To explore the feasibility of electronic PROs (ePRO) collection in recipients ≥65 years old and to compare their compliance to that in recipients 55-64, by evaluating completion rate of the assessment by subjects by age group. | Those completing the assessment at one timepoint 6 months-1 year post-HCT, Those completing the assessment at one timepoint 1 year - 3 years post-HCT, Those completing the assessment at one timepoint Greater than 3 years post-HCT
To identify factors associated with poor compliance with reporting one-time single time ePRO measures in both age groups, by categorizing and quantifying reasons why subjects chose not to participate. | Those completing the assessment at one timepoint 6 months-1 year post-HCT, Those completing the assessment at one timepoint 1 year - 3 years post-HCT, Those completing the assessment at one timepoint Greater than 3 years post-HCT

CONTACTS AND LOCATIONS:
Overall Officials: Bronwen E Shaw, MD, PhD, Principal Investigator — Center for International Blood and Marrow Transplant Research (CIBMTR)/Medical College of Wisconsin
Locations (6):
- United States (6):
  - Stanford University, Stanford, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No